CLINICAL TRIAL: NCT04019249
Title: HealthyWeightHub.fi: Web-based Management of Obesity in a Real-life Clinical Setting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Kirsi Pietiläinen, Professor, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HealthyWeightHub.fi
Record Dates: First submitted 2019-07-12; First posted 2019-07-15 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Obesity
Keywords: eHealth, web-based, internet-based, digital, body weight
MeSH Terms: conditions — Obesity; Body Weight

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Healthy Weight Coaching (Experimental): Intervention: Healthy Weight Coaching.
  Interventions: Behavioral: Healthy Weight Coaching

INTERVENTIONS:
Behavioral: Healthy Weight Coaching — Healthy Weight Coaching is a 52 week long web-based weight loss program consisting of weekly modules, exercises, peer support, and one-on-one coaching. It encompasses themes such as diet, physical activity, coping with stress, sleep, and general health.

SUMMARY:
This study evaluates the effectiveness of a web-based obesity management program HealthyWeightCoaching (HWC), within a HealthyWeightHub.fi (HWH) platform. HWC is a 12-month intervention within a real-life clinical setting. The program includes a combination of nutrition, physical activity, and cognitive behavioral approaches, with a strong basis in acceptance and commitment therapy.

In addition to the automated, interactive program, HWC includes a personal coach allocated to each patient. The patients are enrolled through referrals from primary care, occupational health, other hospitals, or from private health care units nationwide in Finland.

DETAILED DESCRIPTION:
Obesity is one of the major public health problems globally and it increases the risk of many obesity-associated diseases. Treatment of obesity requires long-term interventions, but nevertheless, it is challenging to provide long-term treatment when resources in real-life health care systems are limited. New cost-effective and accessible intervention methods are needed.

The modern treatment of obesity is based on behavioral changes that modify one´s daily lifestyle, which, according to recent research, are effective especially in the prevention of diabetes. However, little is known about the utilization and effectiveness of online programs using novel interactive technologies.

The aim of this study is to evaluate the effectiveness of a real-life web-based obesity management program (HealthyWeightCoaching, HWC) on weight loss, health, quality of life, and factors predicting long term success in treating overweight adult patients.

Healthy Weight Coaching is a novel 12-month intervention within a real-life clinical setting. The program includes a combination of nutrition, physical activity, and cognitive behavioral approaches, with a strong basis in acceptance and commitment therapy. The program is structured around weekly exercise modules.

In addition to the automated, interactive program, HWC includes a personal coach allocated to each patient. The patients are enrolled through referrals from primary care, occupational health, other hospitals, or from private health care units nationwide in Finland. The program is free for the patient to use.

The 12-month intervention is followed by a 5-year monitoring period. Questionnaires on health, quality of life, and lifestyle are collected at 0, 3, 6, 9, and 12-month time points. Body weight is collected by weekly logs. The recruitment is ongoing as the program is currently used in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* body mass index (BMI) ≥ 25 kg/ m²
* the possibility to use a computer and /or a smartphone with access to the internet
* willingness to participate in the digital treatment program

Exclusion Criteria:

* diagnosed severe illness requiring assessment from the specialty care obesity center
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
% weight loss | baseline to 12 months
  Mean weight change in %

SECONDARY OUTCOMES:
Categorical weight loss | baseline to 12 months
  % patients achieving 3-4.9%, 5-9.9% and >10% weight loss
Sleep | baseline to 12 months
  Self-reported sleep variables are measured by a questionnaire that was modified from the Basic Nordic Sleep Questionnaire and The National FINRISK study. Included are questions about sleep duration, chronotype, tiredness, sleep apnoea, and medication.
Health-Related Quality of Life | baseline to 12 months
  Health-related quality of life is measured by the RAND36 questionnaire.
Psychological Flexibility | baseline to 12 months
  Psychological flexibility is assessed by the Acceptance and Action Questionnaire for Weight (AAQW). It is a 22-item, Likert-type scale that measures acceptance of weight related thoughts and feelings with valued actions.
Eating behaviour | baseline to 12 months
  Eating behavior is assessed by the Three Factor Eating Questionnaire (TFEQ), measuring dietary restraint, disinhibition, and susceptibility to hunger.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsi Pietiläinen, MD-PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- University of Helsinki, Helsinki, Finland

REFERENCES:
- [Derived] Mannisto SA, Joki A, Suojanen LU, Venalainen MS, Pietilainen KH, Ahola AJ. Does loneliness impact intentional weight loss? The role of obesity-related disadvantages and comorbidities. Prev Med. 2026 Jan;202:108430. doi: 10.1016/j.ypmed.2025.108430. Epub 2025 Oct 11. PMID 41082943
- [Derived] Ahola AJ, Suojanen LU, Joki A, Pietilainen KH. Loneliness and its cross-sectional associations with health, health behaviours, and perceptions in Finnish patients with overweight or obesity taking part in the Healthy Weight Coaching. Prev Med. 2024 Aug;185:108032. doi: 10.1016/j.ypmed.2024.108032. Epub 2024 Jun 6. PMID 38851400
- [Derived] Biehl A, Venalainen MS, Suojanen LU, Kupila S, Ahola AJ, Pietilainen KH, Elo LL. Development and validation of a weight-loss predictor to assist weight loss management. Sci Rep. 2023 Nov 24;13(1):20661. doi: 10.1038/s41598-023-47930-y. PMID 38001145
- [Derived] Suojanen LU, Ahola AJ, Kupila S, Korpela R, Pietilainen KH. Effectiveness of a web-based real-life weight management program: Study design, methods, and participants' baseline characteristics. Contemp Clin Trials Commun. 2020 Aug 13;19:100638. doi: 10.1016/j.conctc.2020.100638. eCollection 2020 Sep. PMID 32885090
- See also: The HealthyWeightHub portal, into which the HealthyWeightCoaching program is embedded (in Finnish and Swedish only) — https://www.terveyskyla.fi/painonhallinta